CLINICAL TRIAL: NCT03301064
Title: Brief Intervention by Community Health Workers for Unhealthy Drinking in Latinos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of California, San Diego (Other); Providence Health & Services (Other); Boston University (Other)
Responsible Party: Principal Investigator, Mitchell Karno, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-000242
Record Dates: First submitted 2017-09-28; First posted 2017-10-04 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Drinking Heavy; Drinking Behavior; Drinking Excessive
Keywords: alcohol, intervention, Latino, community
MeSH Terms: conditions — Drinking Behavior | interventions — Motivational Interviewing; Ethanol

STUDY DESIGN:
Intervention Model Description: The study is a phase 2 randomized controlled trial to determine the efficacy of a 3-session intervention that combines Motivational Enhancement Therapy and Strengths Based Case Management (MET/SBCM) to reduce unhealthy alcohol use. Participants (n=234) will be block randomized to either the MET/SBCM intervention or to a control condition that receives an educational brochure about alcohol and its associated risks. Both the MET/SBCM intervention and the control condition (i.e., the educational brochure) will be provided by promotores who work for the Providence Center for Community Improvement in Los Angeles, California. Participants will be Latinos served by Providence's outreach programs who exceed low-risk drinking guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition: MET/SBCM (Experimental): The combined Motivational Enhancement Therapy and Strengths Based Case Management (MET/SBCM) intervention will be used in the proposed study. The intervention consists of three 1-hour sessions. The sessions are structured to provide feedback to participants about their risks associated with alcohol use and to help them identify barriers and motivators to change. The sessions will aim to reduce drinking by promoting self-efficacy to change, setting goals and fostering utilization of medical, mental health and social services as needed. A comprehensive list of referrals will be provided. Sessions will occur 1-2 weeks apart.
  Interventions: Behavioral: Motivational Enhancement Therapy and Strengths Based Case Management (MET/SBCM); Other: Alcohol education brochure
- Control Condition: Alcohol education brochure (Active Comparator): Participants randomized to the control condition will be receive a Spanish-language version of an alcohol education brochure. Participants will be encouraged to read the brochure. The brochure will provide information about defining heavy drinking, harmful effects of drinking and symptoms of an alcohol use disorder. Control group participants will also receive a list of available clinics and resources from Providence staff. After the baseline visit participants in the control group will be contacted by phone twice over the next 4 weeks by the promotores to remind them about the 3-month follow-up appointment.
  Interventions: Other: Alcohol education brochure

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy and Strengths Based Case Management (MET/SBCM) — Key objectives of the intervention are as follows: (1) identify health and personal goals and develop discrepancies between goals and current actions, (2) provide feedback related to risks associated with the participant's drinking (e.g., driving after drinking, liver disease), (3) provide normative feedback about the participant's pattern of drinking to alcohol use in the US among Latinos in the participant's age and gender group, (4) discuss reasons for drinking (e.g., feeling isolated from family, machismo, low status employment), (5) weigh the pros and cons of drinking and reasons to reduce drinking (e.g., to better provide for the family, improving family relationships), (6) negotiate a plan for reducing drinking and/or seeking help, (7) recognize personal strengths in the process of change (e.g., religiosity, desire to provide for family), and (8) identify needed social and health services and explore potential barriers (e.g., transportation).
  Arms: Intervention Condition: MET/SBCM
Other: Alcohol education brochure — The alcohol education brochure will address health risks associated with alcohol use and will provide information on low-risk drinking.

SUMMARY:
Latinos will comprise nearly 30% of the population by 2050, and socially disadvantaged Latinos experience a greater burden of poor health and negative social consequences related to their alcohol use than non-Latino Whites. Despite the need for services, low treatment utilization rates and poor treatment retention suggest it is important to make alcohol interventions more accessible for Latinos. Community health workers are an effective way to help under-served populations manage chronic illnesses such as diabetes and hypertension, but they have been used very little in addiction services. The current study extends work from a pilot study that utilized community health workers to deliver a brief alcohol intervention that integrates Motivational Enhancement Therapy and Strengths-Based Case Management (MET/SBCM). Based on those promising but preliminary findings, this study will test the MET/SBCM intervention among a broader population of socially disadvantaged Latinos who engage in unhealthy drinking. For the study a partnership will be formed between the University of California, Los Angeles (UCLA) and a large community-based healthcare organization, Providence Center for Community Health Improvement to conduct a randomized controlled trial of the MET/SBCM intervention.

Participants (n=234) will screen positive for exceeding US low-risk drinking guidelines and will not be seeking alcohol treatment. They will be randomized to either the 3-session MET/SBCM alcohol intervention or to an alcohol brochure control condition. Alcohol use, alcohol-related problems and utilization of health and social services will be assessed at baseline, 3-, and 6-month follow-ups. It is predicted that the MET/SBCM intervention will improve outcomes compared to the control group. The study will also examine the extent to which changes in drinking were preceded by improvements in readiness to change, perceived benefits and risks associated with alcohol use, perception of drinking norms, use of pro-change language during intervention sessions, belief in one's ability to change, self-esteem and use of community services.

The goal of this project is to establish an evidence base for an intervention approach that is sustainable by a large community-based organization serving Latinos. Working with community health workers poises this intervention to address health disparities within this community. The project will help improve the reach and impact of effective alcohol interventions among socially disadvantaged Latinos, thereby contributing to improved population health.

DETAILED DESCRIPTION:
Latinos will comprise nearly 30% of the population by 2050, and socially disadvantaged Latinos experience a greater burden of poor health and negative social consequences related to their alcohol use than non-Latino Whites. The burden of poor health related to alcohol use also suggests the need for early identification and intervention before alcohol use progresses to a more serious condition requiring intensive treatment. Despite the need for services, low treatment utilization rates and poor treatment retention suggest it is important to make alcohol interventions more accessible for Latinos. Spanish-language motivational interventions have been shown to reduce heavy drinking in diverse populations, yet access to these types of interventions remains a limitation. Community health workers are an effective way to help under-served populations manage chronic illnesses such as diabetes and hypertension, but they have been used very little in addiction services. Preliminary evidence from a randomized pilot trial suggested that an intervention integrating Motivational Enhancement Therapy and Strengths Based Case Management (hereafter referred to as MET/SBCM) led to greater reductions in alcohol use compared to a brief feedback condition among socially disadvantaged Spanish speaking Latino male day laborers who were heavy drinkers. Multi-level interventions such as MET/SBCM that target the complex individual- and community-level needs for health-disparities populations are highly recommended as a strategy to improve population health. In that pilot trial the MET/SBCM intervention was provided in Spanish by community health workers (promotores) with high fidelity and participants reported high treatment satisfaction. The results are encouraging for moving forward with additional efforts to study alcohol interventions delivered by community health workers. Based on these promising but preliminary findings, we propose to test the multi-level MET/SBCM intervention targeting a broader population of socially disadvantaged Latinos who engage in unhealthy drinking. For the proposed study a partnership will be formed between UCLA and a large community-based healthcare organization, Providence Center for Community Health Improvement (Providence) to conduct a phase 2 randomized controlled trial. Providence has a well established Latino Health Promoter Program that serves a large population of Latinos, most of whom have low income, low education status and limited English proficiency. The MET-SBCM intervention, to be conducted by promotores at Providence, is thus poised to provide Latinos access to a needed health service for unhealthy alcohol use. If successful, the study will extend the potential reach and impact of brief alcohol intervention for Latinos in the general population.

Primary Aim #1 is to determine the efficacy of the MET/SBCM intervention compared to an educational booklet control condition in reducing alcohol use and alcohol-related problems among Latinos who report exceeding US low-risk drinking guidelines (for men: 5 or more drinks weekly or 15 or more drinks in a given week; for women: 4 or more drinks weekly or 8 or more drinks in a given week).

Hypothesis 1: Participants assigned to a 3-session MET/SBCM intervention will show decreases in the average drinks consumed per week, the frequency of heavy drinking days, and alcohol-related problems at 3- and 6-month follow-ups compared to participants assigned to the educational booklet control condition.

Primary Aim #2 is to determine the efficacy of the MET/SBCM intervention in increasing utilization of community services (e.g., job services, housing assistance, food assistance, mental health services) among Latinos who report exceeding US low-risk drinking guidelines.

Hypothesis 2: Participants assigned to the MET/SBCM intervention will utilize more types of services by the 3- and 6-month follow-ups compared to participants assigned to the educational booklet control condition.

Primary Aim #3 is to examine mechanisms of behavior change underlying observed MET/SBCM intervention effects on alcohol use (or in the event the intervention is not effective, to identify negative findings in the causal chains). Candidate mechanisms are selected based on theory and the extant literature on brief motivation-based interventions and strengths-based case management. The mechanisms will include (1) readiness to change, (2) perceived reward value and risks associated with alcohol use, (3) perception of drinking norms, (4) change talk, (5) general self-efficacy, (6) self-esteem and (7) utilization of community services. We predict that changes in these mechanisms by the 3-month follow-up will mediate the effects of the intervention on average drinks per week at the 6-month follow-up.

The overarching goal of this project is to establish an evidence base for an intervention approach that is ultimately sustainable by a large community-based organization serving Latinos. Working with community health workers positions this intervention to address larger health disparities within this community. The project is significant in its efforts to improve the reach and impact of effective alcohol interventions among socially disadvantaged Latinos, thereby contributing to improved population health.

ELIGIBILITY:
Inclusion Criteria:

* Latino ethnicity
* aged 21 years or older
* speak Spanish (monolingual Spanish or bilingual Spanish and English)
* exceeding low-risk drinking guidelines set by the NIH/NIAAA (for men: 15 or more drinks per week or 5 or more drinks on an occasion weekly in the past month; for women: consuming 8 or more drinks per week or 4 or more drinks on an occasion weekly in the past month)

Exclusion Criteria

* seeking treatment for alcohol problems
* any alcohol treatment in the past 30 days
* serious alcohol withdrawal symptoms as indicated by a score of 10 or higher on the Clinical Institute Withdrawal Assessment for Alcohol-Revised
* substantial problems associated with illicit drug use as indicated by a score of 6 or higher on the Drug Abuse Screening Test (DAST-10)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Percentage of heavy drinking days | 6 months
  Percentage of days on which participants drank heavily in the past 90 days, as defined by NIAAA guidelines (>=5 drinks for men; >=4 drinks for women).

SECONDARY OUTCOMES:
Average number of standard drinks per week | 6 months
  Average number of standard drinks per week in the past 90 days.

OTHER OUTCOMES:
Drinker Inventory of Negative Consequences (DrINC) | 6 months
  Negative consequences associated with alcohol use will include the domains of physical, interpersonal, intrapersonal, impulse control and social responsibility problems. The primary measure of consequences will be the total score across all 5 domains.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell P Karno, PhD, Principal Investigator — University of California, Los Angeles; Alison A Moore, MD, MPH, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - Providence Center for Community Improvement, Van Nuys, California
  - Providence Health and Services, Wilmington, California

IPD SHARING:
Plan to Share IPD: No